CLINICAL TRIAL: NCT01078155
Title: Evaluation of the Role of Adalimumab on Extraarticular Manifestation - Bone Metabolism and Bone Mineral Density in Patients With Active Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-733
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis; Osteoporosis
Keywords: Bone mineral density; Bone turnover markers; Rheumatoid arthritis; Osteoporosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoporosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — osteocalcin (OC), C-terminal type I procollagen peptide (CICP), C-telopeptide of type I collagen (CTX-I), whole blood (serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Active Rheumatoid Arthritis (RA): Participants (women and men) with active early and long-standing RA according to American College of Rheumatology revised criteria from 1987 were prescribed adalimumab in the usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication as well as local guidelines. The decision to prescribe or not to prescribe an anti-TNF was taken prior to a participant's enrollment in the study.

SUMMARY:
This post marketing observational study will be conducted in a prospective, single country, multicenter format to assess the prevention of generalized bone loss in patients with active rheumatoid arthritis (RA) treated with adalimumab (Humira®) in pragmatic prescribing situations. The investigational sites will be centers with experience in the treatment of RA patients and anti-tumor necrosis factor-alpha (TNF-a) therapy. The investigators will be rheumatologists authorized by the Czech Rheumatologic Society for prescribing biological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active early and long-standing RA according to American College of Rheumatology (ACR) 1987 revised criteria.
* Patients with high disease activity DAS28 ≥ 5.1 according to the Czech Rheumatological Society criteria.
* Patients must fulfill national guidelines for use of anti-TNF: inadequate clinical response to at least one disease-modifying antirheumatic drug (DMARD; methotrexate, sulphasalazine, leflunomide, hydroxychloroquine, or combinations) and oral glucocorticoids (equivalent to ≥ 5 mg prednisolone per day), (for Romania except glucocorticoids); chest X-ray, purified protein derivative (PPD)-skin test, Quantiferon/tuberculosis (TB) Gold test (if available) negative for TB.

Exclusion Criteria:

* Patients who have had a history of TNF blocking or rituximab therapy.
* Patients who are being treated or will be treated with drug at risk of interaction with adalimumab (Humira).
* Pregnant females and/or females without adequate method of contraception.
* Patients who didn't receive prior DMARD therapy.
* Patients participating in another study or clinical trial.
* Patients with severe osteoporosis (T-score [number that indicates whether or not bone loss has occurred] of ≤ -2.5 and/or prior vertebral fracture/s).
* Patients with a history of total hip replacement of both extremities.
* Patients who currently receive and/or received bone metabolism modulating agents including Selective Estrogen Receptor Modulators (SERMs), bisphosphonates, parathyroid hormone or anti-receptor activator of nuclear factor-kappaB ligand (RANKL) therapy.
* Subjects who are not eligible for TNF-blocking therapy according to the Czech National Registry (ATTRA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2009-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maroš Lipták, MD, Study Director — Abbvie, Czech Republic & Slovakia

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Active Rheumatoid Arthritis (RA): Participants (women and men) with active early and long-standing RA according to American College of Rheumatology revised criteria from 1987 were prescribed adalimumab in the usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication as well as local guidelines. The decision to prescribe or not to prescribe an anti-tumor necrosis factor (TNF) was taken prior to a participant's enrollment in the study.
Period: Overall Study
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Started | 131
Completed | 87
Not Completed | 44
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 16
Not completed — Participant's Decision | 6
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 123
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD) of Spine and Hip by Dual-energy X-ray Absorptiometry (DEXA) at Baseline, Month 12, and Month 24
Description: BMD of spine and hip (L1-L4 and proximal femur) by DEXA, evaluated according to standard clinical guidelines.
Time Frame: Baseline (Day 0), Month 12, Month 24
Population: Per-Protocol Set: all participants who participated in every study visit; n=participants with evaluable data at time point.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
g/cm^2
  L1-L4 BMD: Baseline; n=86 | 1.06 (0.15)
  L1-L4 BMD: Month 12; n=71 | 1.07 (0.17)
  L1-L4 BMD: Month 24; n=59 | 1.06 (0.17)
  Proximal Femur BMD: Baseline; n=86 | 0.88 (0.14)
  Proximal Femur BMD: Month 12; n=72 | 0.91 (0.13)
  Proximal Femur BMD: Month 24; n=58 | 0.90 (0.13)

2. Primary Outcome: Spine and Hip T-score and Z-score by DEXA at Baseline, Month 12, and Month 24
Description: T-score and Z-score of spine and hip (L1-L4 and proximal femur) by DEXA. T-score is the number of standard deviations that bone density is above or below the average. A score of ≥ -1 = normal bone density; < -1 and > -2.5 = a sign of osteopenia (bone density below normal); ≤ -2.5 = a sign of osteoporosis. Z-score is the number of standard deviations above or below what's normally expected for someone of matching age, sex, weight, and ethnic or racial origin. A Z-score ≤ -2 may suggest abnormal bone loss due to conditions other than aging.
Time Frame: Baseline (Day 0), Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: standard deviations
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
standard deviations
  L1-L4 T-score: Baseline; n=85 | -0.57 (1.14)
  L1-L4 T-score: Month 12; n=71 | -0.42 (1.15)
  L1-L4 T-score: Month 24; n=58 | -0.40 (1.15)
  L1-L4 Z-score: Baseline; n=82 | -0.02 (1.14)
  L1-L4 Z-score: Month 12; n=67 | 0.15 (1.08)
  L1-L4 Z-score: Month 24; n=54 | 0.21 (1.09)
  Proximal Femur T-score: Baseline; n=85 | -0.70 (1.11)
  Proximal Femur T-score: Month 12; n=72 | -0.60 (0.97)
  Proximal Femur T-score: Month 24; n=55 | -0.68 (1.03)
  Proximal Femur Z-score: Baseline; n=82 | -0.18 (1.05)
  Proximal Femur Z-score: Month 12; n=68 | -0.10 (0.96)
  Proximal Femur Z-score: Month 24; n=52 | -0.14 (1.04)

3. Primary Outcome: Change in Bone Turnover Marker Osteocalcin (OC) From Baseline Through Month 3, Month 12, and Month 24
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: Per-Protocol Set: all participants who participated in every study visit; n=participants with bone turnover markers at time point.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
µg/L
  Baseline - Month 3; n=6 | -2.97 (4.68)
  Baseline - Month 12; n=9 | -2.21 (11.99)
  Baseline - Month 24; n=5 | 1.39 (8.77)

4. Primary Outcome: Change in Bone Turnover Marker C-terminal Type I Procollagen Peptide (CICP) From Baseline Through Month 3, Month 12, and Month 24
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
ng/mL
  Baseline - Month 3; n=8 | 8.70 (17.78)
  Baseline - Month 12; n=11 | -1.87 (17.22)
  Baseline - Month 24; n=7 | 15.29 (21.18)

5. Secondary Outcome: Swollen Joint Count at Baseline, Month 3, Month 12, and Month 24
Description: The investigator counted the number of swollen joints at each study visit (28 joints are routinely examined).
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
joints
  Baseline; n=87 | 9.5 (4.91)
  Month 3; n=87 | 2.3 (2.76)
  Month 12; n=87 | 1.0 (1.57)
  Month 24; n=84 | 1.0 (1.22)

6. Secondary Outcome: Disease Activity Score in 28 Joints (DAS28) at Baseline, Month 3, Month 12, Month 24
Description: Scores on the DAS28 range from 0 to 10. DAS 28 ≥ 5.1= high RA disease activity; DAS 28 ≥ 3.2 = middle RA disease activity; DAS 28 ≤ 3.2 = lower disease activity; DAS 28 ≤ 2.6 = remission of disease.
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
units on a scale
  Baseline; n=87 | 6.24 (0.73)
  Month 3; n=87 | 3.55 (1.13)
  Month 12; n=85 | 2.86 (1.04)
  Month 24; n=75 | 2.83 (0.93)

7. Secondary Outcome: Visual Analogue Scale (VAS): Physician's Global Assessment of Disease Activity at Baseline, Month 3, Month 12, Month 24
Description: Physician's Global Assessment of Disease Activity VAS was reported on a 100 mm scale, where 0 = very good to 100 = very bad.
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: Per-Protocol Set: all participants who participated in every study visit, with evaluable data at time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 86
units on a scale
  Baseline | 68.0 (11.77)
  Month 3 | 29.7 (16.69)
  Month 12 | 23.0 (15.50)
  Month 24 | 21.5 (13.45)

8. Primary Outcome: Change in Bone Turnover Marker C-telopeptide of Type I Collagen (CTX-I) From Baseline Through Month 3, Month 12, and Month 24
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
µg/L
  Baseline - Month 3; n=14 | -0.01 (0.09)
  Baseline - Month 12; n=14 | 0.06 (0.46)
  Baseline - Month 24; n=11 | -0.01 (0.28)

9. Primary Outcome: Mean Duration of Morning Stiffness at Baseline, Month 3, Month 12, and Month 24
Description: Participant-reported the existence and duration of morning stiffness, defined as "morning stiffness in and around the joints, lasting at least 1 hour before maximal improvement."
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
minutes
  Baseline; n=84 | 95.0 (58.34)
  Month 3; n=60 | 37.5 (42.48)
  Month 12; n=51 | 27.7 (34.63)
  Month 24; n=53 | 25.8 (27.27)

10. Primary Outcome: Tender Joint Count at Baseline, Month 3, Month 12, and Month 24
Description: The investigator counted the number of tender joints at each study visit (28 joints are routinely examined).
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
joints
  Baseline; n=87 | 14.3 (6.52)
  Month 3; n=87 | 3.1 (3.01)
  Month 12; n=87 | 1.9 (2.39)
  Month 24; n=84 | 1.7 (1.88)

11. Secondary Outcome: Visual Analogue Scale (VAS): Subject's Global Assessment of Disease Activity at Baseline, Month 3, Month 12, Month 24
Description: Subject's Global Assessment of Disease Activity VAS was reported on a 100 mm scale, reporting the subject's evaluation of his/her difficulties as 0 = without any difficulty to 100 = significant difficulties.
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
units on a scale
  Baseline; n=86 | 71.1 (12.36)
  Month 3; n=86 | 31.4 (16.18)
  Month 12; n=85 | 24.7 (15.18)
  Month 24; n=85 | 24.0 (14.37)

12. Secondary Outcome: Visual Analogue Scale (VAS): Subject's Assessment of Pain at Baseline, Month 3, Month 12, Month 24
Description: Subject's Assessment of Pain VAS was reported on a 100 mm scale, where 0 = no pain through 100 = severe pain.
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
units on a scale
  Baseline; n=86 | 71.3 (12.38)
  Month 3; n=86 | 29.4 (14.33)
  Month 12; n=85 | 25.8 (16.56)
  Month 24; n=85 | 24.2 (15.51)

13. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) at Baseline, Month 3, Month 12, Month 24
Description: ESR was recorded as per local clinical practice. Normal findings are up to 20 mm/hr for females and up to 15 mm/hr for males.
Time Frame: Baseline (Day 0), Month 3, Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/1 hour
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 87
mm/1 hour
  Baseline; n=65 | 37.77 (21.06)
  Month 3; n=64 | 17.97 (14.91)
  Month 12; n=65 | 17.15 (14.13)
  Month 24; n=63 | 17.67 (12.34)

ADVERSE EVENTS:
Time Frame: 268 weeks and 5 days (adverse event and serious adverse event analyses did not include those cases where the onset followed the last dose of study drug for > 70 days).
Arm/Group | Participants With Active Rheumatoid Arthritis (RA)
Serious Adverse Events (participants affected / at risk) | 1/131
Other Adverse Events (participants affected / at risk) | 11/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Active Rheumatoid Arthritis (RA) (N=131)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Active Rheumatoid Arthritis (RA) (N=131)
Dermatitis Allergic (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Cutaneous Vasculitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.